CLINICAL TRIAL: NCT05679739
Title: NEUROprotection Via optimizINg Cerebral Blood Flow afTer cArdiaC arresT (NEURO-INTACT) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEURO-INTACT
Record Dates: First submitted 2022-10-30; First posted 2023-01-11 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest (OHCA)
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized blood pressure strategy (Experimental): Hemodynamic optimization performed to an individualized target mean arterial pressure in the first 72 hours post ROSC based on cerebral perfusion assessed serially.
  Interventions: Other: Individualized blood pressure strategy

INTERVENTIONS:
Other: Individualized blood pressure strategy — An individualized blood pressure strategy targeting cerebral blood flow, serially guided by near-infrared spectroscopy and transcranial Doppler ultrasound. Assessments are performed on admission, and at 12, 24 and 48 hours post-ROSC.

SUMMARY:
This single-center proof of concept study aims to assess the efficacy of a blood pressure strategy targeting person- and time-specific cerebral blood flow compared with standard-of-care using neuron-specific enolase as a quantitative biomarker of brain injury. Our central hypothesis is that an individualized blood pressure strategy targeting cerebral perfusion will reduce the extent of brain injury as indicated by changes in levels of neuron-specific enolase from baseline at 72 hours. To test this hypothesis, we will recruit 49 patients to an individualized blood pressure management strategy targeting cerebral blood flow, where optimal blood pressure will be serially calculated by the ICM+ brain monitoring software (Cambridge, UK) using inputs from transcranial Doppler ultrasound and near-infrared spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. At least 21 years of age
2. Comatose defined as not being able to obey verbal commands and no verbal response to pain after sustained ROSC.

Exclusion Criteria:

1. ≥ 80 years old at time of enrolment
2. Pregnant patients
3. Limitations of care or life support therapy withdrawn within 24 hours of admission

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mean change in neuron-specific enolase (NSE) | 72 hours post ROSC
  The mean change in concentration of NSE from baseline levels to 72 hours post-ROSC.

SECONDARY OUTCOMES:
Peak concentration of myocardial injury biomarker - High-sensitive troponin (hsTNT) | Within 72hours of ROSC
  Peak concentration of myocardial injury biomarker, High-sensitive troponin (hsTNT) within 72 hours of ROSC
Peak concentration of myocardial injury biomarker - N-terminal pro b-type natriuretic peptide (NT-proBNP) | Within 72hours of ROSC
  Peak concentration of myocardial injury biomarker, N-terminal pro b-type natriuretic peptide (NT-proBNP) within 72 hours of ROSC
Peak concentration of renal function - Creatinine | Within 72hours of ROSC
  Peak concentration of renal function, Creatinine within 72 hours of ROSC
Peak concentration of renal injury biomarker - Proenkephalin A 119-159 (penKID) | Within 72hours of ROSC
  Peak concentration of renal injury biomarker, Proenkephalin A 119-159 (penKID) within 72 hours of ROSC
Peak concentration of renal injury biomarker - Biologically active adrenomedullin (bio-ADM) | Within 72hours of ROSC
  Peak concentration of renal injury biomarker, Biologically active adrenomedullin (bio-ADM) within 72 hours of ROSC
Peak concentration of renal injury biomarker - Tissue inhibitor of metalloproteinases 2 (TIMP2) | Within 72hours of ROSC
  Peak concentration of renal injury biomarker, Tissue inhibitor of metalloproteinases 2 (TIMP2) within 72 hours of ROSC
Peak concentration of renal injury biomarker - Insulin Like Growth Factor Binding Protein 7 (IGFBP7) | Within 72hours of ROSC
  Peak concentration of renal injury biomarker, Insulin Like Growth Factor Binding Protein 7 (IGFBP7) within 72 hours of ROSC
Neurological outcome | Through study completion, average of 12 months post OHCA
  Neurological outcomes measured by Cerebral Performance Category (CPC) scale on hospital discharge, and at 3, 6 and 12 months post OHCA. The CPC purports to assess domains of functioning after cardiopulmonary resuscitation (CPR) with scores ranging from 1 (good cerebral performance/normal life) to 5 (brain death).
Physical function | Through study completion, average of 12 months post OHCA
  Physical function measured by the change of Duke Activity Status Index (DASI) self-reported questionnaire on hospital discharge, and at 3, 6 and 12 months post OHCA. DASI score is the sum of the questionnaire responses, score of 34 or less means moderate-to-severe complications.
Neurocognitive outcome - Montreal Cognitive Assessment (MOCA) | Through study completion, average of 12 months post OHCA
  Neurocognitive is assessed by Montreal Cognitive Assessment (MOCA, global cognition) on hospital discharge, and at 3, 6 and 12 months post OHCA. Scores on the MOCA from zero to 30, while score of 26 and above is considered normal.
Neuropsychological outcome - Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Through study completion, average of 12 months post OHCA
  Neuropsychological deficits is assessed by the modified local version of Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) on hospital discharge, and at 3, 6 and 12 months post OHCA. Standard scores of 70 and above will classify as average/mild impairment, scores 55 to 69 as moderate impairment and severe impairment for scores less than 55.
Neuropsychological outcome- Depression, Anxiety, and Stress Scale (DASS-21) | Through study completion, average of 12 months post OHCA
  Depression, Anxiety, and Stress Scale (DASS-21) is used to assess neuropsychological outcome on hospital discharge, and at 3, 6 and 12 months post OHCA.
Health-related quality of life | Through study completion, average of 12 months post OHCA
  Health-related quality of life measured by EuroQol-5 Dimension-5 Level (EQ-5D-5L) questionnaire on hospital discharge, and at 3, 6 and 12 months post OHCA. EQ-5D-5L questionnaire consists of 5 dimensions (mobility, self care, usual activities, pain/comfort, anxiety/depression). There are 5 levels in each dimensions. The lowest level means normal which the highest level means extremely severe.

OTHER OUTCOMES:
Exploratory outcome - Digital neurocognitive assessment | Through study completion, average of 12 months post OHCA
  Neurocognitive is assessed by digital neurocognitive assessment on hospital discharge, and at 3, 6 and 12 months post OHCA.

CONTACTS AND LOCATIONS:
Overall Officials: Shir Lynn Lim, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Heart Centre, Singapore, Singapore, Singapore